CLINICAL TRIAL: NCT00370422
Title: Bevacizumab Versus Combined Bevacizumab and Triamcinolone for Refractory Diabetic Macular Edema; a Randomized Clinical Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8412
Record Dates: First submitted 2006-08-30; First posted 2006-08-31 (Estimated); Last update posted 2007-03-13 (Estimated); Status verified 2005-10

CONDITIONS: Diabetic Macular Edema
Keywords: Cystoid macular edema; Diabetic macular edema; Hard exudates; Intravitreal bevacizumab; Intravitreal triamcinolone; Macular thickness
MeSH Terms: conditions — Macular Edema | interventions — Triamcinolone; Bevacizumab

INTERVENTIONS:
Drug: Triamcinolone, Bevacizumab

SUMMARY:
The purpose of this study is to compare the efficacy and safety of intravitreal injection of bevacizumab alone versus bevacizumab combined with triamcinolone for treatment of refractory diabetic macular edema.

DETAILED DESCRIPTION:
According to the early treatment diabetic retinopathy study (ETDRS), the treatment of choice for diabetic macular edema is laser therapy, which may be neither effective nor curative in some patients. Corticosteroids may have a beneficial effect on diabetic macular edema. Other newly introduced medications for macular edematous lesions are anti-VEGF vascular endothelial growth factor)drugs. In this randomized, sham-controlled, multicenter, three-arm clinical trial,we try to evaluate the safety and efficacy of intravitreal bevacizumab alone and in combination with intravitreal triamcinolone in the treatment of refractory diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Cases with clinically significant macular edema (CSME) with persistent retinal thickening after initial or supplemental macular photocoagulation

Exclusion Criteria:

* Monocularity,
* History of vitrectomy,
* Glaucoma or ocular hypertension,
* Significant media opacity,
* Existence of traction on the macula

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-11; Study Completion 2006-09

PRIMARY OUTCOMES:
Visual acuity
Central macular thickness

SECONDARY OUTCOMES:
Cataract progression
Intraocular pressure
Anterior chamber reaction

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Ahmadieh, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Hamid Ahmadieh, MD, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Ahmadieh H, Ramezani A, Shoeibi N, Bijanzadeh B, Tabatabaei A, Azarmina M, Soheilian M, Keshavarzi G, Mohebbi MR. Intravitreal bevacizumab with or without triamcinolone for refractory diabetic macular edema; a placebo-controlled, randomized clinical trial. Graefes Arch Clin Exp Ophthalmol. 2008 Apr;246(4):483-9. doi: 10.1007/s00417-007-0688-0. Epub 2007 Oct 5. PMID 17917738